CLINICAL TRIAL: NCT05967962
Title: Sensory Modulation Dysfunction as a Risk Factor for Posttraumatic Stress Disorder - A Randomized Control Trial
Brief Title: Sensory Modulation Dysfunction and Posttraumatic Stress Disorder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Tami Bar-Shalita, Principal Investigator, Tel Aviv University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 0005364-2
Record Dates: First submitted 2023-04-08; First posted 2023-08-01 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Posttraumatic Stress Disorder; Sensory Processing Disorder
Keywords: sensory processing; executive function; trauma; peritrauma
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Wounds and Injuries | interventions — Motion Pictures

STUDY DESIGN:
Intervention Model Description: A randomized controlled trial with an experimental group and a control group: Specifically participants will be screened for SMD, thereafter randomization will be applied within each group: with and without SMD, separately.
Who Masked: Outcomes Assessor
Masking Description: Assessors will be blind to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- traumatic (scenes of injury and death during combat) (Experimental): In the experimental group participants will be exposed to a traumatic scene, to simulate combat exposure by watching 16 min traumatic combat scenes from the TV series "When Heroes Fly.
  Interventions: Behavioral: The Trauma Film Paradigm
- non-traumatic (neutral) film (Active Comparator): In this active control group, participants will be watching 16 min. non-traumatic, neutral scene showing combatants as well (scenes from the YouTube series "Warriors").
  Interventions: Behavioral: non-traumatic (neutral) film

INTERVENTIONS:
Behavioral: The Trauma Film Paradigm — Trauma film paradigm is a well-known, validated and established procedure that produces reactions similar to those generated by trauma, and that is often used in research to predict susceptibility for peritraumatic and posttraumatic reactions. In this study the trauma film paradigm will be utilized to simulate combat exposure. The two groups of participants will undergo the trauma film paradigm by watching 16 min traumatic combat scenes vs. non-traumatic movie scenes, respectively. Participants will be given standardized instructions (i.e., ''Imagine you are present at the scene"; "Do not close your eyes").
  Arms: traumatic (scenes of injury and death during combat)
Behavioral: non-traumatic (neutral) film — non-traumatic (neutral) film
  Arms: non-traumatic (neutral) film

SUMMARY:
To explore the role of sensory modulation dysfunction (SMD) (i.e., a neurodevelopmental state altering the sensory perception, severely interfering with daily function) as a risk factor for posttraumatic stress disorder (PTSD), its co-occurring pain, and impeded cognitive functions, following exposure to combat trauma.

DETAILED DESCRIPTION:
Background and Aim: Posttraumatic stress disorder (PTSD) is interwoven with chronic pain, and the latter co-occurs with sensory modulation dysfunction (SMD). Moreover, SMD was found as a risk factor for chronic pain and hampered executive functioning. Currently, the sensory domain is neglected in the PTSD research realm, though findings indicate its link to PTSD. Thus, this study proposes to bridge a current gap in PTSD knowledge base, and specifically, our general aim is to uncover the role of SMD in predicting combat trauma-related symptomatology, altered executive function, and clinical pain.

Methods: This is a single-blind randomized control study, comprising 4 assessments: pre (T1); post (T2); 10 (T3); and 40 (T4) days follow-up, following experimental manipulation (see Figure 1). Participants with and without SMD will be randomly allocated to experimental and control groups that will watch traumatic movie scenes simulating combat and non-traumatic movie scenes, respectively. The assessor will be blinded to group allocation.

Population: One-hundred healthy individuals aged 18 to 28 years, with and without SMD. Participants with SMD will be identified via a standardized questionnaire during screening. The sample size was calculated based on power analyses via G*Power 3 software derived from p-value of .05 and statistical power of .80.

Tools: Both objective and subjective outcome measures will be applied consisting of self-report questionnaires, psychophysical-, physiological-, emotional reactions, and executive function performance-based- testing will be applied. The experimental manipulation will comprise of the Trauma film paradigm.

Expected Results: Findings may advance the understanding of PTSD development and thus not only serve in attenuating the risk for PTSD among combatants but also may contribute to developing preventative measures for PTSD among combatants.

ELIGIBILITY:
Inclusion Criteria:

* Intact or corrected vision
* Proficiency in Hebrew
* Exclusion Criteria:
* Neurological disorders
* Psychiatric disorders
* Neurodevelopmental disorders
* Substance use disorder
* Chronic pain
* Regular intake of medications.
* Cultural and societal backgrounds that might bias participant reaction to study protocol (i.e., nationality)

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-07-30 (Actual); Primary Completion 2024-08-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain Sensitivity Questionnaire (PSQ) | Change from immediately before and immediately after the manipulation and 40 days post undertaking the manipulation
  A 17 item self-report questionnaire assessing daily pain sensitivity, aimed to quantify everyday somatosensory pain sensitivity to imagined painful daily life situations. Participants rate the intensity of imagined pain on a 10-point scale: 'not painful at all' (0) to 'the worst pain imaginable' (10). The Pain Sensitivity Questionnaire provides a total score (range 17-170) and two sub-scores.
Spontaneously occurring memories | Change between T2, T3, T4: SpecificallyT2-during 6 days, starting the day after undertaking the experiment = trauma film paradigm, 10 (T3); and 40 (T4) days follow-up, following experimental manipulation
  Diaries will be utilized for reporting spontaneously occurring memories of the film, consisting of 6 items of which 1 is an open question. This will be filled once a day for 6 days starting the next day after the trauma film paradigm was undertaken. Thereafter, it will be filled in again in T3 and T4

SECONDARY OUTCOMES:
Salivary cortisol | Change between T1 and T2: (immediately before and immediately after the manipulation = trauma film paradigm)
  Using commercially available cortisol electrochemiluminescent immunoassays (ECLIA) kits (Roche Diagnostics GmbH, Mannheim, Germany) on a cobas e801 module (Roche Diagnostics GmbH)
Heart rate | Change between: immediately before (T1) and immediately after the manipulation = trauma film paradigm (T2)
  Recorded via the Mindware BioNex 8-slot chassis acquisition system (Mindware Technologies Ltd, Gahanna,OH, USA
skin conductance | Change between: immediately before (T1) and immediately after the manipulation = trauma film paradigm (T2)
  Recorded via the Mindware BioNex 8-slot chassis acquisition system (Mindware Technologies Ltd, Gahanna,OH, USA
Executive function | Change between T1 and T2: ( immediately before and immediately after the manipulation= trauma film paradigm)
  The executive function will be measured using 2 performance-based tests, both testing the same outcomes, to avoid the learning effect which may occur when using one in short intervals: (i) Trail making test (TMT) (at pre-experimental manipulation) and (ii). Color trail test (CTT) (at post-experimental manipulation), alternating between subjects. Both tests are widely used to assess executive function and specifically target visual scanning, processing speed, and capacity to maintain focus attention/mental flexibility, providing 2 scores: speed of completion and error rate.
Quantitative sensory testing- pain psychophysics | Change between T1 and T2: (immediately before and immediately after the manipulation = trauma film paradigm)
  Thermal and pain thresholds using the Thermal Sensory Analyzer (TSA) (Medoc, Israel). The tests will include cold detection threshold (CDT), warm detection threshold (WDT), cold pain threshold CPT) and warm pain threshold (CPT). The TSA thermod's active area is 32 cm and temperature range is 0°C to a safety limit of 50°C. Each test will be performed three times in the dorsal aspects of the dominant hand. Conditioned pain modulation (CPM) will be tested utilizing heat test stimuli individually tailored rated as 50/100, delivered via the TSA thermod to the volar aspect of the dominant hand, conditioned by the contralateral hand immersed in painfully cold water (7C).
Face reading | Change between immediately before (T1) and immediately after the manipulation = trauma film paradigm (T2)
  Utilizing the FaceReader hardware (incl.: Webcam, LED ring) and the FaceReader software Base module, during the trauma film paradigm manipulation, all participants will be videotaped using the webcam on their computer screen. The videotapes will be analyzed offline using the FaceReader software Base module to classify emotional reactions
The State- Trait anxiety Inventory (STAI) | Change between T1 and T2: (immediately before and immediately after the manipulation= trauma film paradigm)
  A self-report 2 part questionnaire, assessing both anxiety state and anxiety trait, comprising 20 items each. All items are rated on a 4-point scale (e.g., from "Almost Never" to "Almost Always"). Higher scores indicate greater anxiety. In this study, only the Anxiety state part will be utilized
Dissociation-Tension-Scale | T2: (immediately after the manipulation= trauma film paradigm)
  A 21-item self-report questionnaire designed to assess psychological and somatoform dissociative features. Ratings are made on a 10-point scale ranging from 0 (not at all) to 9 (very much).
Distress after trauma film paradigm | T2: (immediately after the manipulation= trauma film paradigm)
  Three questions self-report aiming at rating participant experience due to the movie scene: 2 with a response scale of 1 ("not distressed") to 10 ("extremely distressed"), and one with a response scale of 1 ( very pleasant) to 5 (very unpleasant), constructed for the purpose of this current study
The Impact of Event Scale-Revised (IES-R) | Change between T3 and T4: (10 and 40 days post undertaking the manipulation =trauma film paradigm)
  Self-report questionnaire for testing Trauma-related symptomatology. The IES-R comprises 22 items that measure symptoms of intrusion (dreams about the event), avoidance and numbing (the effort to avoid reminders of the event), and hyperarousal (feeling watchful and on guard) with respect to a potentially traumatic event. Participants are asked to rate on a 5-point Likert scale the extent to which each item applies to their experiences. The total score on the IES-R ranges between 0 and 88.
Skin conductance | Change between: immediately before (T1) and immediately after (T2) the manipulation = trauma film paradigm)
  Recorded via the Mindware BioNex 8-slot chassis acquisition system (Mindware Technologies Ltd, Gahanna,OH, USA

OTHER OUTCOMES:
Sensory responsiveness questionnaire (SRQ) | Baseline ( screening phase)
  A 58-item questionnaire aimed at clinically classifying sensory modulation dysfunction in adults. Items represent typical daily life situations involving auditory, visual, gustatory, olfactory, vestibular and somatosensory sensations, excluding pain. Items are phrased either in a hedonic or aversive valence and are graded on a 5-point Likert scale: 'not at all' (1) to 'very much' (5). Two cut-off scores are provided. Will be used for group allocation: Individuals with vs. without sensory modulation dysfunction. As mentioned in study design trauma film paradigm randomization will be applied within each of these groups separately.
The Dissociation Experiences Scale-II (DES-II) | Baseline ( screening phase)
  A 28-item self-report questionnaire that measures the frequency of dissociative experiences. The total dissociative score was computed as the mean of these 28 items, ranging from 0 to 100.
Vividness of Visual Imagery Questionnaire (VVIQ) | Baseline ( screening phase)
  A 16-question instrument assessing visual imagery. Participants are asked to imagine a number of specified items determined by the test protocol and to rate their subjective impression of vividness on a Likert scale ranging from 1 (perfectly clear and as vivid as normal vision) to 5 (no image at all, you only " know" that you are thinking of the object).
Life Events Checklist for DSM-5 (LEC-5) | Baseline ( screening phase)
  It is a 17-item self-report measure assessing lifetime potentially traumatic event types. Participants rate each item with six response options: happened to me, witnessed it, learned about it, part of my job, not sure, or doesn't apply.
Post Traumatic Groth Inventory (PTGI) | Baseline ( screening phase)
  A self-report scale assessing posttraumatic growth consisting of 21 statements. Participants are asked to rate the extent to which the indicated change occurred in their lives as a result of their stressful/traumatic life experiences" Each item was scored on a 4-point scale ranging from 1 (I didn't experience this change at all) to 4 (I experienced this change to a very great).
PTSD Checklist for DSM-5 (PCL-5) | Baseline ( screening phase)
  In this 20-item self-report measure, assessing subclinical PTSD symptoms, participants are asked to indicate the extent to which they experienced each PTSD symptom, on a 5-point Likert scale ranging from 0 (not at all) to 4 (extremely). Items corresponded to the newly approved PTSD symptom criteria in the Diagnostic and Statistical Manual of Mental Disorders. In this study will be used for screening
Difficulties in Emotion Regulation Scale (DERS) | Baseline ( screening phase)
  A 16-item self-report questionnaire designed to assess individuals' typical levels of emotion dysregulation. Participants are asked to rate the extent to which each item applies to them on a 5-point Likert-type scale from 1 (almost never) to 5 (almost always).

CONTACTS AND LOCATIONS:
Overall Officials: Tami Bar-Shalita, PhD, Principal Investigator — Tel Aviv University; Yael Lahav, PhD, Principal Investigator — Tel Aviv University; Michal Lifshitz, MD, Principal Investigator — Israel Defense Forces
Locations (1):
- Dr. Tami Bar-Shalita, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No
Will be available upon request